CLINICAL TRIAL: NCT02416089
Title: Tampostat: A Low-cost, Self-regulating Tamponade for Management of Postpartum Hemorrhage in Bangladesh
Brief Title: Tampostat for Management of Postpartum Hemorrhage
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Grand Challenges Canada (Other); Jibon Health Technologies, Inc. (Industry); Shaheed Suhrawardi Medical College Hospital (Unknown); Dhaka Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-14095
Record Dates: First submitted 2015-03-16; First posted 2015-04-14 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2016-11

CONDITIONS: Postpartum Hemorrhage
Keywords: Tampostat; Tamponade; Postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tampostat (Experimental): Tampostat™ is a self-regulating, low cost, pressure based emergency obstetric device designed specifically for use in low-resource settings. It has 6 parts: probe, condom, O ring, nerve centre, tube and bulb pump. It offers significant benefits over the current model by simplifying the insertion process, reducing the need for constant monitoring, eliminating leakage and the need for sterile saline, and using a pressure-based mechanism to apply consistent pressure to all women regardless of uterus size.Women who develop PPH even after applying AMTSL at the hospital or women who visit the hospital with PPH within 24 hours after delivery will be managed by Tampostat for the intervention arm or by the condom catheter tamponade in the control arm(172 patients in each arm)
  Interventions: Device: Tampostat
- Condom catheter tamponade (Active Comparator): Condom catheter tamponade have been used by medical professionals for several years in the management of atonic (primary) PPH. In this approach, Sterile rubber catheter fitted with a condom as a tamponade balloon device and using normal saline to inflate the condom.
  Interventions: Device: Condom catheter tamponade

INTERVENTIONS:
Device: Tampostat
  Arms: Tampostat
Device: Condom catheter tamponade
  Arms: Condom catheter tamponade

SUMMARY:
The purpose of the study is to evaluate the safety, feasibility and applicability of a new device 'Tampostat' in the management of primary postpartum hemorrhage and compare the efficacy of 'Tampostat' in terms of arresting primary PPH with that of the conventional condom catheter.

DETAILED DESCRIPTION:
This will be a 2-year study having two parts. Part A will be a Proof of Concept (POC) study that will be conducted at the Obstetrical Ward of Shaheed Suhrawardi Medical College Hospital (ShSMCH) and Dhaka Medical College Hospital (DMCH). There is no sample size estimation of this POC study that will assess safety, feasibility and applicability of using Tampostat on 5 consenting women with PPH for each hospital. Part B of the study will be an open label, randomized clinical trial that will be conducted at the Obstetrical Ward of Dhaka Medical College Hospital (DMCH). In this part, 344 consenting women with primary PPH will be enrolled, and allocated to either Tampostat or the control intervention in equal numbers per randomization (172 patients in each arm). In both these parts, Tampostat will be used only when Active Management of Third Stage of Labour (AMTSL) has failed to prevent PPH within 24 hours after delivery. All the doctors involved in the provision of care and treatment to PPH patients will be trained on the WHO's standard of care; they will also receive training on appropriate use of the devices to be used in this trial. An expert committee constituted of OBGYN professionals, clinical trial specialists, and statisticians will oversee the technical management of patients, data collection and their procedures, and ethical issues in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Women who delivered their baby at the site hospital, or attended the site hospital with PPH that started within the last 24 hours.
2. Women with primary PPH have received AMTSL.
3. PPH is due to atonic uterus.
4. Provides written informed consent for enrolment in the study.

Exclusion Criteria:

1. Primary PPH caused by retained placenta or ruptured uterus.
2. Women who delivered before 28 weeks of gestation.
3. Women not willing to participate in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Safety of Tampostat as measured by number of serious adverse events in primary PPH management | 2 months
  The safety of Tampostat [no. of Serious adverse events i.e. Incidence of air embolism, injury to the uterine wall, pain during inflation of condom & continuation of vaginal /uterine bleeding during use of Tampostat] in primary PPH management.
Efficacy of Tampostat as measured by number of successful cases in arresting bleeding in Primary PPH | 12 months
  Efficacy [number of successful cases in arresting bleeding due to primary PPH from atonic uterus] of Tampostat in the management of primary postpartum hemorrhage (PPH)
Comparison of the efficacy of Tampostat as measured by number of successful cases in arresting primary PPH and the time takes to arrest the bleeding with that of the condom catheter tamponade | 12 months
  Comparison of the efficacy of Tampostat in terms of arresting primary PPH due to atonic uterus with that of the conventional condom catheter tamponade [no. of successful cases in arresting primary post partum bleeding using Tampostat and condom catheter and the time both takes to arrest the bleeding]

SECONDARY OUTCOMES:
Feasibility as measured by number of physicians consider Tampostat as a feasible device in arresting primary PPH | 2 months
  The feasibility of Tampostat[number of physicians consider Tampostat as a feasible device in arresting primary PPH due to atonic uterus] in the management of primary PPH by
Applicability of Tampostat as measured by rating by service providers using pre established scoring system in the management of primary PPH | 2 months
  Applicability[rating by service providers on applicability of the device using pre established scoring system]of Tampostat in the management of primary PPH due to atonic uterus.

CONTACTS AND LOCATIONS:
Overall Officials: Aminur Rahman, MBBS,MSc, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Obstetrical Ward of Shaheed Suhrawardi Medical College Hospital (ShSMCH) and Dhaka Medical College Hospital (DMCH), Dhaka, Bangladesh

REFERENCES:
- [Background] Condous GS, Arulkumaran S, Symonds I, Chapman R, Sinha A, Razvi K. The "tamponade test" in the management of massive postpartum hemorrhage. Obstet Gynecol. 2003 Apr;101(4):767-72. doi: 10.1016/s0029-7844(03)00046-2. PMID 12681884
- [Background] Vitthala S, Tsoumpou I, Anjum ZK, Aziz NA. Use of Bakri balloon in post-partum haemorrhage: a series of 15 cases. Aust N Z J Obstet Gynaecol. 2009 Apr;49(2):191-4. doi: 10.1111/j.1479-828X.2009.00968.x. PMID 19432609
- [Result] Seligman, B. and X. Liu, Economic assessment of interventions for reducing postpartum hemorrhage in developing countries. 2006: Abt Associates.
- [Result] Organization, W.H., Make Every Mother and Child Count: The World Health Report. 2005: World Health Organization.
- [Result] Khan KS, Wojdyla D, Say L, Gulmezoglu AM, Van Look PF. WHO analysis of causes of maternal death: a systematic review. Lancet. 2006 Apr 1;367(9516):1066-1074. doi: 10.1016/S0140-6736(06)68397-9. PMID 16581405
- [Result] National Institute of Population Research and Training (NIPORT), M.E., and icddr,b, Bangladesh Maternal Mortality and Health Care Survey 2010, M.E. NIPORT, and icddr,b, Editor. 2012: Dhaka.
- [Result] Lalonde A, Daviss BA, Acosta A, Herschderfer K. Postpartum hemorrhage today: ICM/FIGO initiative 2004-2006. Int J Gynaecol Obstet. 2006 Sep;94(3):243-53. doi: 10.1016/j.ijgo.2006.04.016. Epub 2006 Jul 12. PMID 16842791
- [Result] Prendiville WJ, Elbourne D, McDonald S. Active versus expectant management in the third stage of labour. Cochrane Database Syst Rev. 2000;(3):CD000007. doi: 10.1002/14651858.CD000007. PMID 10908457
- [Result] Abu-Heija AT, Jallad FF. Emergency peripartum hysterectomy at the Princess Badeea Teaching Hospital in north Jordan. J Obstet Gynaecol Res. 1999 Jun;25(3):193-5. doi: 10.1111/j.1447-0756.1999.tb01146.x. PMID 10467792
- [Result] Bakri YN, Amri A, Abdul Jabbar F. Tamponade-balloon for obstetrical bleeding. Int J Gynaecol Obstet. 2001 Aug;74(2):139-42. doi: 10.1016/s0020-7292(01)00395-2. PMID 11502292
- [Result] Doumouchtsis SK, Papageorghiou AT, Arulkumaran S. Systematic review of conservative management of postpartum hemorrhage: what to do when medical treatment fails. Obstet Gynecol Surv. 2007 Aug;62(8):540-7. doi: 10.1097/01.ogx.0000271137.81361.93. PMID 17634155
- [Result] Georgiou C. Balloon tamponade in the management of postpartum haemorrhage: a review. BJOG. 2009 May;116(6):748-57. doi: 10.1111/j.1471-0528.2009.02113.x. PMID 19432563
- [Result] Seror J, Allouche C, Elhaik S. Use of Sengstaken-Blakemore tube in massive postpartum hemorrhage: a series of 17 cases. Acta Obstet Gynecol Scand. 2005 Jul;84(7):660-4. doi: 10.1111/j.0001-6349.2005.00713.x. PMID 15954876
- [Result] Rather, S.Y., et al., Use of condom to control intractable PPH. JK science, 2010. 12(3)
- [Result] Rathore AM, Gupta S, Manaktala U, Gupta S, Dubey C, Khan M. Uterine tamponade using condom catheter balloon in the management of non-traumatic postpartum hemorrhage. J Obstet Gynaecol Res. 2012 Sep;38(9):1162-7. doi: 10.1111/j.1447-0756.2011.01843.x. Epub 2012 Apr 30. PMID 22540529
- [Result] Tindell K, Garfinkel R, Abu-Haydar E, Ahn R, Burke TF, Conn K, Eckardt M. Uterine balloon tamponade for the treatment of postpartum haemorrhage in resource-poor settings: a systematic review. BJOG. 2013 Jan;120(1):5-14. doi: 10.1111/j.1471-0528.2012.03454.x. Epub 2012 Aug 13. PMID 22882240
- [Result] Georgiou C. Intraluminal pressure readings during the establishment of a positive 'tamponade test' in the management of postpartum haemorrhage. BJOG. 2010 Feb;117(3):295-303. doi: 10.1111/j.1471-0528.2009.02436.x. Epub 2009 Nov 26. PMID 19943825
- [Result] Mirski MA, Lele AV, Fitzsimmons L, Toung TJ. Diagnosis and treatment of vascular air embolism. Anesthesiology. 2007 Jan;106(1):164-77. doi: 10.1097/00000542-200701000-00026. PMID 17197859
- [Result] Shaikh N, Ummunisa F. Acute management of vascular air embolism. J Emerg Trauma Shock. 2009 Sep;2(3):180-5. doi: 10.4103/0974-2700.55330. PMID 20009308
- [Result] Akhter S, Begum MR, Kabir Z, Rashid M, Laila TR, Zabeen F. Use of a condom to control massive postpartum hemorrhage. MedGenMed. 2003 Sep 11;5(3):38. PMID 14600674
- [Derived] Kellie FJ, Wandabwa JN, Mousa HA, Weeks AD. Mechanical and surgical interventions for treating primary postpartum haemorrhage. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013663. doi: 10.1002/14651858.CD013663. PMID 32609374